CLINICAL TRIAL: NCT01013506
Title: A Phase II Trial of Endocrine Therapy in Combination With OSI-906 (an IGF-1R Inhibitor) With or Without Erlotinib (Tarceva, an EGFR Inhibitor) in Patients With Hormone-sensitive Metastatic Breast Cancer.
Brief Title: Phase 2, Endocrine Therapy + OSI-906 With or Without Erlotinib for Hormone-sensitive Metastatic Breast Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was abandoned before opening to accrual. Replaced by another study.
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Ingrid Mayer, MD, Assistant Professor of Medicine; Clinical Director, Breast Cancer Program; Medical Oncologist, Vanderbilt-Ingram Cancer Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VICC BRE 0977; P30CA068485 (NIH); VU-VICC-BRE-0977
Record Dates: First submitted 2009-11-12; First posted 2009-11-13 (Estimated); Last update posted 2013-05-23 (Estimated); Status verified 2013-05

CONDITIONS: Breast Cancer
Keywords: estrogen receptor-positive breast cancer; progesterone receptor-positive breast cancer; stage IV breast cancer; recurrent breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — 3-(8-amino-1-(2-phenylquinolin-7-yl)imidazo(1,5-a)pyrazin-3-yl)-1-methylcyclobutanol; Erlotinib Hydrochloride; Goserelin; Letrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Letrozole +/-goserelin, OSI-906 (Arm I ) (Experimental): Patients receive oral letrozole once daily on days 1-28 plus subcutaneous goserelin (the latter for pre-menopausal women only) on day 1 and oral IGF-1R inhibitor OSI-906 twice daily on days 1-28. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: IGF-1R inhibitor OSI-906; Drug: goserelin; Drug: letrozole
- Letrozole +/- goserelin, OSI-906, erlotinib (Arm II) (Experimental): Patients receive oral letrozole and subcutaneous goserelin (the latter for pre-menopausal women only) and oral IGF-1R inhibitor OSI-906 as in arm I. Patients also receive oral erlotinib hydrochloride once daily on days 1-28. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: IGF-1R inhibitor OSI-906; Drug: erlotinib hydrochloride; Drug: goserelin; Drug: letrozole

INTERVENTIONS:
Drug: IGF-1R inhibitor OSI-906 — Given orally
Drug: erlotinib hydrochloride — Given orally
  Other Names: Tarceva
  Arms: Letrozole +/- goserelin, OSI-906, erlotinib (Arm II)
Drug: goserelin — Given subcutaneously
  Other Names: Zoladex
Drug: letrozole — Given orally
  Other Names: Femara

SUMMARY:
RATIONALE: Estrogen can cause the growth of breast cancer cells. Hormone therapy using letrozole +/- goserelin (the latter for pre-menopausal women only) may fight breast cancer by lowering the amount of estrogen the body makes. OSI-906 and erlotinib hydrochloride may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. It is not yet known whether hormone therapy and OSI-906 are more effective when given with or without erlotinib hydrochloride in treating hormone-sensitive metastatic breast cancer.

PURPOSE: This phase II trial is studying how well giving hormone therapy together with OSI-906 with or without erlotinib hydrochloride works in treating hormone-sensitive patients with metastatic breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the antitumor activity of letrozole +/- goserelin (the latter for pre-menopausal women only) in combination with IGF-1R inhibitor OSI-906 with or without erlotinib hydrochloride, measured by time to progression, in patients with hormone-sensitive metastatic breast cancer.

Secondary

* To determine the safety of these regimens in these patients.
* To determine the response rate in patients treated with these regimens.
* To measure circulating C-peptide, IGF-1, and IGFBP-3 levels in patients treated with these regimens.
* To correlate the expression of IGF-IR, EGFR, HER2, Y1316 and Y1131 pIGF-1R, PTEN, S473 pAkt, pMAPK, S118 (MAPK site), and S167 (Akt and S6 site) pER in formalin-fixed paraffin blocks (FFPB) with clinical outcome and luminal A vs. luminal B subtypes of breast cancer.
* To correlate the mutational status of PI3K (E542K, E545K, H1047R) in DNA extracted from FFPB or fresh biopsy with clinical outcome and luminal A vs. luminal B subtypes of breast cancer

OUTLINE: This is a multicenter study. Stratification will be based on previous exposure to endocrine therapy: (Arm I) no previous endocrine therapy or have completed adjuvant therapy > 6 months prior to study enrollment; (Arm II) patients that had previous endocrine therapy in the metastatic setting or had metastatic recurrence within 6 months of adjuvant endocrine therapy.

* Arm I: Patients receive oral letrozole once daily on days 1-28 +/- subcutaneous goserelin* on day 1 and oral IGF-1R inhibitor OSI-906 twice daily on days 1-28. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.
* Arm II: Patients receive oral letrozole +/- subcutaneous goserelin* and IGF-1R inhibitor OSI-906 as in arm I. Patients also receive oral erlotinib hydrochloride once daily on days 1-28. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.

NOTE: *Goserelin will only be given to premenopausal patients.

Tumor tissue samples from original diagnosis or from fresh biopsy tissue are collected for biomarker analysis and other studies.

After completion of study therapy, patients are followed periodically.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed invasive breast carcinoma

  * Stage IV disease
* No locally recurrent resectable disease
* No symptomatic brain metastases

  * History of brain metastases allowed provided the patient is clinically stable for > 3 weeks after completion of radiotherapy AND is not taking steroids or therapeutic anticonvulsants that are CYP3A4 modifiers
* Hormone receptor status:

  * Estrogen receptor and/or progesterone receptor positive tumor by immunohistochemistry (IHC)

PATIENT CHARACTERISTICS:

* Pre- or post-menopausal
* ECOG performance status 0-1
* Life expectancy ≥ 6 months
* ANC ≥ 1,250/mm^3
* Platelet count ≥ 100,000/mm^3
* Creatinine ≤ 1.5 times upper limit of normal (ULN)
* Bilirubin ≤ 1.5 times ULN (≤ 3 times ULN if liver metastasis is present)

  * For patients with Gilbert syndrome, direct bilirubin will be measured instead of total bilirubin
* SGOT and SGPT ≤ 1.5 times ULN (≤ 3 times ULN if liver metastasis is present)
* Alkaline phosphatase ≤ 1.5 times ULN (≤ 3 times ULN if liver metastasis is present)
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective barrier contraception during and for 3 months after completion of study therapy
* Able to swallow and retain oral medication
* Baseline QTc ≤ 450 msec
* No other invasive cancer within the past 5 years except for completely resected basal cell or squamous cell skin cancer or successfully treated cervical carcinoma in situ
* No malabsorption syndrome significantly affecting gastrointestinal function
* No diabetes, fasting glucose > 150mg/dL, or receiving ongoing anti-hyperglycemic therapies
* No concurrent uncontrolled illness including, but not limited to, any of the following:

  * Ongoing or active infection requiring parenteral antibiotics
  * Impaired lung function (i.e., COPD or lung conditions requiring oxygen therapy)
  * Symptomatic congestive heart failure (NYHA class III or IV heart disease)
  * Unstable angina pectoris, angioplasty, stenting, or myocardial infarction within the past 6 months
  * Uncontrolled hypertension, defined as systolic BP > 180 mm Hg or diastolic BP > 100 mm Hg on two consecutive measurements taken ≥ 1 week apart, despite adequate medical support
  * Clinically significant cardiac arrhythmia (multifocal premature ventricular contractions, bigeminy, trigeminy, or ventricular tachycardia that is symptomatic or requires treatment)
  * Psychiatric illness and/or social situation that would compromise patient safety or limit compliance with study requirements, including maintenance of a compliance/pill diary

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Recovered from prior therapy
* At least 2 weeks since prior investigational drugs
* No more than 4 prior chemotherapy treatments in the metastatic setting

  * Does not include endocrine therapy or single-agent biologic therapy
* No concurrent CYP3A4 or CYP1A2 modifiers
* No other concurrent anticancer therapy, including chemotherapy, radiotherapy, surgery, immunotherapy, hormonal therapy, or biologic therapy

  * Concurrent radiotherapy to painful bone metastases or areas of impeding bone fracture allowed provided radiotherapy is initiated before study therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-08; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Time to progression | from study entry to date of progressive disease
  Duration from study enrollment to date of progressive disease (PD) as measured by Response Evaluation in Solid Tumors (RECIST) criteria v. 1.1: measurable lesions: PD is > 20% increase in the sum of the longest diameter of target lesions or appearance of new lesions

SECONDARY OUTCOMES:
Safety profile of OSI-906 and letrozole +/ goserelin, with and without erlotinib | at 4 weeks
  The number of patients with worst-grade toxicity at each of five grades following NCI Common Toxicity Criteria: 1 = mild, 2 = moderate, 3 = severe, 4 = life-threatening, disabling, 5 = death
Response | every 12 weeks to progression
  Per RECIST criteria v. 1.1: measurable lesions: complete response (CR) disappearance of target lesions, partial response (PR) > 30% decrease in the sum of the longest diameter (LD) of target lesions, progressive disease (PD) > 20% increase in the sum of the LD of target lesions or appearance of new lesions, stable disease (SD) neither sufficient decrease nor increase of the sum of smallest sum of the LD of target lesions
Circulating C-peptide, IGF-1 | At baseline and on day 1 of each 28-day cycle
  Levels of the protein C-peptide and the hormone IGF-1 in the blood
Correlation of IGF-IR, EGFR, HER2, Y1316 and Y1131 pIGF-1R, PTEN, S473 pAkt, pMAPK, S118 (MAPK site), and S167 (Akt and S6 site) pER expression with time to progression and molecular classification | On receipt of breast tissue: tissue block from prevous surgery or fresh tissue from current surgery
  The levels of these biomarkers will be measured in breast tumor tissue and compared and contrasted with patient's time to progression and molecular classification (luminal A vs. luminal B)
Mutation analysis of PI3K (E542K, E545K, H1047R) | On receipt of breast tissue: tissue block from prevous surgery or fresh tissue from current surgery
  Breast tumor tissue will be examined for mutations in these genes.

CONTACTS AND LOCATIONS:
Overall Officials: Ingrid Mayer, MD, Principal Investigator — Vanderbilt-Ingram Cancer Center